CLINICAL TRIAL: NCT01604512
Title: Enhancing Brain Lesions After Radiation Therapy: A Comparison of MRI Perfusion and FDG PET/CT to Distinguish Between Radiation Injury and Tumor Progression
Brief Title: A Comparison of MRI Perfusion and FDG PET/CT to Distinguish Between Radiation Injury and Tumor Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-067
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-02

CONDITIONS: Brain Cancer
Keywords: Brain tumor; MRI Perfusion; FDG PET/CT; 12-067
MeSH Terms: conditions — Brain Neoplasms | interventions — Perfusion Magnetic Resonance Imaging; Positron Emission Tomography Computed Tomography

ARMS (1):
- Pts with a brain tumor (Experimental): The study will prospectively enroll patients who have increasing size and/or enhancement of brain lesion(s) after brain radiation therapy for a neoplasm (either primary or metastatic), where. it is unclear if a lesion represents radiation injury or progressive tumor. At the discretion of PI the RSI sequence may be repeated at SOC FDG or other radiotracer imaging carried out while the patient is still on study, if deemed clinically necessary.
  Interventions: Diagnostic Test: MRI perfusion and PET/CT scans

INTERVENTIONS:
Diagnostic Test: MRI perfusion and PET/CT scans — The MRI perfusion and PET/CT scans will be obtained within 12 weeks of each other. These scans are part of the standard of care for patients with brain tumors and uncertain tumor response or progression after treatment. Although every effort will be made to perform both MRI perfusion and PET/CT on the same day or during the same week, some patients may experience longer intervals between scans due to scheduling conflicts. The disease in question (radiation injury vs. tumor progression) may change slightly during this interval (e.g., the lesion may grow or shrink slightly), but no large changes are expected between the two scans. The patients may continue existing treatments in the interval between scans (e.g., steroids, chemotherapy), but the two scans must be performed before any change or new treatment occurs. Fusion images of MRI and PET/CT will not be reviewed by the neuroradiologist interpreting the MRI perfusion nor the nuclear medicine radiologist interpreting the PET/CT.

SUMMARY:
This study will examine if MRI perfusion and PET/CT can tell growing tumor and radiation injury apart. MRI perfusion looks at the blood vessels in the tumor. PET/CT looks if the tumor cells are actively growing. The investigators will do these two tests and see which one is better.

Patients will remain on study until the completion of either the MRI perfusion or PET/CT that are within 12 weeks of each other. After one of these scans, the patient will have no active interventions and will be off study.

Optional: Restriction Spectrum Imaging (RSI) Sequence RSI sequence is an advanced way of looking at your brain. The scan allows doctors to see how water is moving within brain tumors or within brain cells. The extra sequence takes additional 4-5 minutes in the scanner. The RSI sequence is optional. The patient will only be asked to participate if the doctor believes that it will be helpful.

Off study: Patients will remain on study until the completion of either the MRI perfusion or PET/CT that are within 12 weeks of each other. After one of these scans, the patient will have no active interventions and will be off study. Patients will obtain a standard of care brain MRI scan about every 2-3 months. These MRI scans will be used to track disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Pathological or clinical/radiological diagnosis of aneoplasm , either primary (e.g., malignant glioma) or secondary (metastasis from systemic malignancy) with a history of brain radiation therapy
* Completed fractionated radiation therapy (to 60 Gy for high grade gliomas) or stereotactic radiosurgery or hypofractionated radiation therapy (e.g. for brain metastases, anaplastic meningiomas), without or with concurrent chemotherapy
* New or increased enhancing brain lesion(s) OR nonenhancing brain lesion(s) if receiving anti-angiogenic therapy, which is considered indeterminate for tumor progression vs. radiation injury by the neuroradiologist or clinician
* Patient and/or guardian is able to provide written informed consent prior to study registration
* Age ≥ 18 years old

Exclusion Criteria:

* Claustrophobia
* Known allergic reaction to Gd-DTPA
* Any contraindication to gadolinium intravenous contrast as per standard Department of Radiology contrast guidelines
* Any contraindication to MRI (e.g., pacemaker, aneurysm clip, tissue expander).
* Pregnant or nursing female
* Unable to cooperate for MRI and/or PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-05; Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Young, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pts With a Brain Tumor
Started | 148
Completed | 141
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Not treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pts With a Brain Tumor
Number analyzed (Participants) | 148
Age, Continuous [Median (Full Range); unit: years] | 56 [20 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 124
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received PET/CT and MRI Perfusion Studies
Description: To assess the utility of PET/CT and MRI perfusion studies in predicting whether worsening enhancing brain lesions seen after radiation therapy represent radiation injury or tumor progression. This study will examine the role of these two imaging techniques in predicting diagnosis and treatment planning.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With a Brain Tumor
Number analyzed (Participants) | 148
Participants
  Participants who received PET/CT and MRI perfusion studies | 53
  Participants who did not receive PET/CT and MRI perfusion studies | 95

2. Secondary Outcome: Median Time Between Radiation Therapy and Detection of Indeterminate Lesion
Description: Median time between Radiation Therapy and detection of indeterminate lesion
Time Frame: up to 99 months
Measure: Median (Full Range); unit: months
Arm/Group | Pts With a Brain Tumor
Number analyzed (Participants) | 148
months | 9 [1 to 99]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pts With a Brain Tumor
All-Cause Mortality (participants affected / at risk) | 18/148
Serious Adverse Events (participants affected / at risk) | 6/148
Other Adverse Events (participants affected / at risk) | 0/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With a Brain Tumor (N=148)
Death NOS (General disorders) | 5
Seizure (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT01604512/Prot_SAP_000.pdf